CLINICAL TRIAL: NCT00398944
Title: Impact of a Computerized Decision Support System, Based on EBM French Guidelines, on the Management of Hypertension and Diabetes: a Randomised Controlled Trial in Primary Care
Brief Title: Impact of a Computerized Guidelines on the Management of Hypertension and Diabetes
Acronym: ASTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société de Formation Thérapeutique du Généraliste (Other)
Responsible Party: Doctor Hector Falcoff, Société de Formation Thérapeutique du Généraliste
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SFTG1968A
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2006-11

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: Guideline based decision support system, Hypertension, Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Evaluation of the impact of a guideline based computerized decision support system.

SUMMARY:
The purpose is to determine wether an electronic decision support system based on national guidelines is effective to improve the follow-up and the treatment of two conditions: hypertension and diabetes, in primary care practices.

DETAILED DESCRIPTION:
Existing computer-based ordering systems for physicians provide drug-centred checks but offer little assistance for optimizing the overall patient-centred treatment strategy.

The ASTI project aims :

1. to design a guideline-based decision support system for diabetic and/or hypertensive patients, to help general practitioners :

   1. to carry out procedures (clinical and biological tests) according to guidelines (the recommended procedure at the recommended moment), and to get a synthetic view of all the elements they need to follow-up the patient
   2. to avoid prescription errors and to improve compliance with therapeutic guidelines. The " critic mode " operates as a background process and corrects the physician's prescription on the basis of automatically triggered elementary rules that account for isolated guideline recommendations. The " guided mode " directs the physician to the best treatment by browsing a comprehensive guideline knowledge base represented as a decision tree.
2. To measure the impact of ASTI when it is implemented with an electronic medical record system. We adopt a randomized design, with the practice as the unit of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension
* Mellitus diabetes
* Follow-up by GP's

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2715 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Patients who underwent the recommended procedures during the last 12 months | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Hector FALCOFF, Principal Investigator — Société de Formation Thérapeutique du Généraliste
Locations (1):
- SFTG, Paris, France

REFERENCES:
- [Background] Seroussi B, Bouaud J, Dreau H, Falcoff H, Riou C, Joubert M, Simon C, Simon G, Venot A. ASTI: a guideline-based drug-ordering system for primary care. Stud Health Technol Inform. 2001;84(Pt 1):528-32. PMID 11604796